CLINICAL TRIAL: NCT04830254
Title: Correlation Between Selected Hematological and Doppler Ultrasonic Parameters After Electrical Stimulation in Peripheral Arterial Diseased Patients
Brief Title: Correlation Between Selected Haematological and Doppler Ultrasonic Parameters in Peripheral Arterial Diseased Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TENS21
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group(A) (Active Comparator): Group (A) included 20 patients who received low-frequency TENS (frequency 4 Hz, pulse duration 200 μs) for 45 min per session, three times per week, and for 12 weeks.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation(TENS) device
- Control group(B) (Sham Comparator): The control group(B) included 20 patients who received placebo TENS stimulation but with a voltage level falling to zero after 10 s of stimulation
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation(TENS) device

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation(TENS) device — The Patients in group (A) received low-frequency TENS (frequency 4 Hz, pulse duration 200 μs,burst mode) was be applied through 2 output channels surface electrodes with an E2 TENS device, for 45 min per session, supramaximal stimulation to sympathetic ganglions in T12, L1, and L2, which innervate the lower extremity . For 45 min per session, three times per week, and for 12 weeks.
  Other Names: TENS

SUMMARY:
Forty patients of both sexes, aged between 50 and 60 years, were chosen from an outpatient vascular clinic in the El Sahel Education Hospital. Patients have been examined and referred to by a vascular specialist.

DETAILED DESCRIPTION:
The participants were divided randomly into two groups of equal numbers. The study group got low-frequency TENS (4 Hz frequency, pulse duration 200 μs) which was administered through surface electrodes for 45 min per session, supramaximal stimulation for T12, L1, and L2 sympathetic ganglions that innervate the lower extremity for 45 min per session, three times per week and for 12 weeks. Control Group that received placebo stimulation as provided by the same TENS device but with a zero volt after 10 s of stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral Leriche-Fontaine stage-II PAD
2. Both sexes
3. Aged 50 to 60 years
4. Outpatients
5. Clinically stable
6. Sedentary
7. Not participating in any physical activity last 3 months

Exclusion Criteria:

1. Walking disorders related to orthopedic or neuromuscular disease
2. Renal insufficiency requiring dialysis (Renal diseases)
3. Known and documented myopathy
4. Progressive cancer
5. Associated progressive disease causing a deterioration in general health
6. Participation in another research protocol
7. Skin disorder making it impossible to use TENS
8. Absolute contraindication to physical activity
9. Presence of a pacemaker/defibrillator

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Red cell distribution width (RDW) | change from baseline to after 12 weeks
  Peripheral venous blood samples were obtained from each patient.
Mean platelet volume(MPV) | change from baseline to after 12 weeks
  Peripheral venous blood samples were obtained from each patient.
Ankle peak systolic velocity (APSV) | change from baseline to after 12 weeks
  is the mean of the peak systolic velocities of the anterior and posterior tibial arteries measured at the ankle level by doppler ultrasonography
Arterial diameter | change from baseline to after 12 weeks
  Diameter of lower limb arteries measured by doppler ultrasonography

SECONDARY OUTCOMES:
Actual claudication distance | change from baseline to after 12 weeks
  Claudication pain distance was measured after running on a treadmill constant walking speed of 2 mile/hour at 0% grade, with gradual increases in grade of 2.0% every 2 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No